CLINICAL TRIAL: NCT05333315
Title: The Effects of Five Different Food Supplements With Restriction Diet on the Components of the Metabolic Syndrome in Overweight and Obese Adults
Brief Title: Clinical Trials of Five Different Food Supplements With Restriction Diet in Adults
Acronym: FOODSU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Biostile d.o.o. (Unknown)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate professor, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Food supplements_CLINICAL
Record Dates: First submitted 2022-04-01; First posted 2022-04-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Overweight and Obesity; Inflammation; Hypercholesterolemia; Hypertension
Keywords: food supplements; diet; metabolic syndrome
MeSH Terms: conditions — Overweight; Obesity; Inflammation; Hypercholesterolemia; Hypertension; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Investigation Product 1 (IP1) in softchews form (Experimental): 0,5 g of glucomannan per softchew
  Interventions: Dietary Supplement: IP1
- Investigation Product 2 (IP2) in powder form (Experimental): Fiber of light Indian plantain, 7 g; glucomannan, 4,3 g; Inulin 2,5 g; Apple fiber, 1g; Choline, bitartrate 90 mg; Apple pectin,50 mg; Inositol, 40 mg
  Interventions: Dietary Supplement: IP2
- Investigation Product 3 (IP3) in powder form and capsules form (Experimental): POWDER: Plantain fibre 10 g; Inulin, 2 g; Apple fibre, 1,5 g; Root of pellitory, 500 mg; Apple pectin, 450 mg CAPSULE: Pumpkin seed extract, 300 mg; Garlic extract odourless, 300 mg; Artichoke leaf extract, 150 mg; Cumin seed extract, 150 mg; Peppermint leaf extract, 150 mg; Anise seed extract, 150 mg; Curcuma rhizome extract, 150 mg; Vitamin C, 42 mg; Zinc (in gluconate),10 mg; Vitamin B6, 1,5 mg
  Interventions: Dietary Supplement: IP3
- Investigation Product 4 (IP4) in liquid form (Experimental): LIQUID: Arabinogalactan, 700 mg; Inulin, 700 mg; Beta-glucans, 30 mg
  Interventions: Dietary Supplement: IP4
- Investigation Product 5 (IP5) in two capsules form (Experimental): CAPSULE 1:L-arginine, 100 mg; Choline bitartrate, 100 mg; L-carnosine, 100 mg; L-taurine, 100 mg; Soy lecithin, 50 mg; R-alfa lipoic acid,10 mg; Vitamin B6,2 mg; Folic acid, 200 µg; Vitamin D3, 5 µg; Vitamin B12, 2 µg CAPSULE 2: Schisandra fruit extract, 400 mg; Milk thistle fruit extract associated with phospholipids, 200 mg; Grape seed extract associated with phospholipids, 50 mg; Grape seed extract (Vitis vinifera),50 mg
  Interventions: Dietary Supplement: IP5

INTERVENTIONS:
Dietary Supplement: IP1 — IP1: 2 softchews 3 times a day before meals with 1-2 glasses of water for eight weeks.
  OTHER: Placebo
  Arms: Investigation Product 1 (IP1) in softchews form
Dietary Supplement: IP2 — IP2: One bag per day mixed in 200 mL of cold water or tea and consumed immediately, on an empty stomach, half an hour before breakfast for eight weeks.
  OTHER: Placebo
  Arms: Investigation Product 2 (IP2) in powder form
Dietary Supplement: IP3 — IP3: One bag per day in the morning, dissolved in a glass of warm water and three capsules per day with a glass of water or tea (one capsule at breakfast, one at lunch and one at dinner) for eight weeks.
  OTHER:Placebo
  Arms: Investigation Product 3 (IP3) in powder form and capsules form
Dietary Supplement: IP4 — IP4: Twice a day 20 mL half an hour before breakfast and half an hour before dinner for eight weeks.
  OTHER:Placebo
  Arms: Investigation Product 4 (IP4) in liquid form
Dietary Supplement: IP5 — IP5: Formula 1: One capsule per day at breakfast with a glass of water for eight weeks and Formula 2: Two capsules a day at breakfast and at dinner with a glass of water for eight weeks.
  OTHER:Placebo
  Arms: Investigation Product 5 (IP5) in two capsules form

SUMMARY:
In recent years, dietary supplement are of great interest for the improvement of human health. This study is designed as a parallel, randomized, double blind study exploring the efficacy of two months daily oral dosing of five different food supplements together with diet restriction in 120 otherwise healthy overweight or obese adults on different biochemical and anthropometric parameters.

DETAILED DESCRIPTION:
The incidence of obesity has been rapidly increasing, and this condition has become a major public health threat, since it is strongly linked with increased risk for several diseases including type 2 diabetes, cardiovascular disease, cancer and brain aging. Obesity and overweight are chronic disorders of multifactorial origin that are characterized by high oxidative status and by low chronic inflammation. Thus far, molecular mechanisms underlying obesity and obesity-related metabolic disorders have not been fully clarified, and effective therapeutic approaches to lower inflammation and oxidative stress are currently of general interest.

In recent years, dietary supplement and are of interest for the improvement of human health. This study is designed as a parallel, randomized, double blind study exploring the efficacy of two months daily oral dosing of five different food supplements together with diet restriction in 120 otherwise healthy overweight or obese adults on different biochemical (lipid profile, glucose, C-reactive protein, bilirubin, alanine aminotransferase, etc), and anthropometric parameters (body mass, the percentage of body fat, visceral fat index, etc,...). Food supplements are mainly composed of different fiber and other bioactive compounds.

ELIGIBILITY:
Inclusion Criteria: BMI > 25 kg/m2

* BMI > 25 kg/m2
* personally signed and dated informed consent form
* ability to understand and willingness to comply with all protocols required visits assessments and interventions

Exclusion Criteria:

* use of dietary supplements
* use of medication for any component of metabolic syndrome
* presence of inflammatory and/or autoimmune disorders
* pregnancy or lactating

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in body fat | eight weeks
  Changes in percentage of body fat from baseline to week eight measured with bioelectrical impedance analysis (BIA) Tanita MC-980MA

SECONDARY OUTCOMES:
Change in body weight | eight weeks
  Changes in body weight (in kilograms) from baseline to week eight measured with bioelectrical impedance analysis (BIA) Tanita MC-980MA
Changes in waist circumference | eight weeks
  Changes in waist circumference (in centimetres) from baseline to week eight measured with a flexible tape measure
Changes in muscle mass | eight weeks
  Changes in muscle mass (in kilograms) from baseline to week eight measured with bioelectrical bioelectrical impedance analysis (BIA) Tanita MC-980MA
Changes in visceral fat rating | eight weeks
  Changes in visceral fat rating (index) from baseline to week eight measured with bioelectrical bioelectrical impedance analysis (BIA) Tanita MC-980MA
Lipid profile | eight weeks
  Changes in total cholesterol, LDL cholesterol, HDL cholesterol and triacylglycerides measured by biochemical analyzer Cobass
Blood pressure | eight weeks
  Changes in diastolic and systolic blood pressure measured by blood pressure device (Omron M3)
Inflammation | eight weeks
  Changes in C-reactive protein levels measured by biochemical analyzer Cobass
Antioxidative potential | eight weeks
  Changes in antioxidative potential determined by 1,1-diphenyl-2-picrylhydrazyl (DPPH) radical measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided